CLINICAL TRIAL: NCT04237870
Title: A Clinical Study to Explore the Effect of Repetitive Transcranial Magnetic Stimulation on Abnormal Executive Function of High Function Autism Spectrum Disorder Children
Brief Title: Effect of rTMS on the Abnormal Executive Function of ASD Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XH-19-013
Record Dates: First submitted 2020-01-19; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Executive Dysfunction; ASD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment (Active Comparator): Active cTBS treatment will be delivered at an intensity that is 70% of the resting motor threshold (RMT). cTBS consist of bursts of 3 magnetic pulses at 30 Hz repeating every 200 ms for 300 pulses. cTBS repeat twice with 15 min interval. Treatment will be applied in central suleus.
  Interventions: Device: Active cTBS
- Sham treatment (Sham Comparator): Sham rTMS will be delivered using the same stimulation parameters and at the site of active treatment, but with only the side-edge resting on the scalp. The coil will be angled 45 degrees way from the skull in a single-wing tilt position. This method produces sound and some somatic sensation (e.g. contraction of scalp muscles) similar to those of active stimulation, but with minimal direct brain effects.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Active cTBS — Active cTBS treatment will be delivered at an intensity that is 70% of the resting motor threshold (RMT). cTBS consist of bursts of 3 magnetic pulses at 30 Hz repeating every 200 ms for 300 pulses. cTBS will be repeated twice with 15 min interval. The cTBS sessions last for 4 weeks, 5 times a week. Treatment will be applied to central suleus.
  Other Names: magstim Rapid2 (Magstim Company Ltd. UK)
  Arms: Active treatment
Device: Sham — Sham stimulation will be delivered using the same stimulation parameters and at the site of active treatment, but with only the side-edge resting on the scalp. The coil will be angled 45 degrees way from the skull in a single-wing tilt position. This method produces sound and some somatic sensation (e.g. contraction of scalp muscles) similar to those of active stimulation, but with minimal direct brain effects.
  Other Names: magstim Rapid2 (Magstim Company Ltd. UK)
  Arms: Sham treatment

SUMMARY:
In this study, the investigators will explore the effects of repetitive transcranial magnetic stimulation (rTMS) on executive function deficits in high function autism spectrum disorder. Half of the participants will be chosen by chance to receive continuous theta burst stimulation (cTBS) while the other half will be chosen by chance to receive sham stimulation. And finally the sham group individuals also receive cTBS. Based on results from a recent unpublished pilot data, the investigators propose that cTBS treatment will induce a significant improvement in executive function performance compared to sham treatment.

DETAILED DESCRIPTION:
This study is a randomized, sham controlled study to evaluate the efficacy of cTBS as a treatment for executive function deficits in individuals with autism spectrum disorder between 6 and 16 years of age. The study duration is approximately 1 months, with the cTBS sessions lasting for 4 weeks, 5 times a week, for about 20min each. Several scales will be used to assess for symptom severity and adaptive functioning. The executive function will be evaluated by Behaviour Rating Inventory of Executive Functioning (BRIEF) questionnaire. Cognition will be assessed using functional near - infrared spectroscopy (fNIRS).

This study also involves a type of brain imaging known as magnetic resonance imaging (MRI) at the beginning and at the end of the 4 weeks daily cTBS to better understand the effects of cTBS on brain structure and function. Investigators will measure the size and connections of different parts of the brain to assess brain structure and blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ASD. Diagnostic criteria: diagnosed by pediatric psychiatrists in accordance with the criteria in the Fifth Edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-V), Autism Diagnostic Observation Schedule (ADOS) and Autism Diagnostic Interview-Revised (ADI-R);
* Have a diagnosis of high functioning ASD (HF-ASD) (i.e., are verbal with an Intelligence Quotient (IQ) ≥ 70)
* Are clinically stable as determined by their treating physician, with no medication changes over the past 4 weeks

Exclusion Criteria:

* Have metal or electronic instruments near the stimulation brain area of coil, such as, have intravascular stent in head, have metal objects in skull.
* Have cardiac pacemaker, cochlear implant, medical pump;
* Can not cooperate with examiner;
* Have intracranial foreign bodies by craniotomy, or intracranial deformity
* Have a history of substance abuse or dependence in the last 6 months or have a positive urine toxicology screen
* Have a concomitant major medical or neurologic illness
* Have had a seizure in the past, or have a first-degree relative with epilepsy
* Have an abnormal clinical EEG
* Are pregnant or likely to get pregnant during the next 4 weeks
* Have a history of rTMS treatment.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in scores on Behaviour Rating Inventory of Executive Functioning (BRIEF) | Baseline; Post cTBS (4 weeks after baseline
  Specifically the investigators will evaluate the changes in executive function (EF) scores before and after cTBS treatment.

SECONDARY OUTCOMES:
Change in scores, reaction time and brain blood flow on the Working Memory Task by fNIRS | Baseline; Post cTBS (4 weeks after baseline)
  Specifically the investigators will evaluate the changes in spatial working memory scores, reaction time and brain blood flow before and after cTBS treatment.
Change in size and connections of different parts of the brain to assess brain structure and blood flow by functional magnetic resonance imaging (fMRI) | Baseline; Post cTBS (4 weeks after baseline)
  Specifically the investigators will evaluate the change in size and connections of different parts of the brain to assess brain structure and blood flow by fMRI before and after cTBS treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Li, PhD, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Fei Li, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No